CLINICAL TRIAL: NCT04692974
Title: Cognitive Frailty in Older Adults: Protocol of a Pilot RCT of the Role of Technology in Physical Activity Enhancement
Brief Title: Cognitive Frailty in Older Adults: The Role of Technology in Physical Activity Enhancement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Sengkang General Hospital (Other)
Responsible Party: Principal Investigator, Rathi Mahendran, Associate Professor, Senior Consultant Psychiatrist, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-20-038
Record Dates: First submitted 2020-12-10; First posted 2021-01-05 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Mild Cognitive Impairment; Frailty
Keywords: Cognitive Frailty; Physical Frailty; Physical Activity; Mild Cognitive Impairment; Technology
MeSH Terms: conditions — Cognitive Dysfunction; Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention and control group design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization will be carried out by a research assistant not involved in the study.
  The assessors will be blind to the treatment assignment of the participant when administering the questionnaires.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will be given the wearables which they will use together with the accompanying mobile application for the period of the study (6 months). During the period of intervention, the wearable will track the physical activity of the older adults via the number of steps taken and number of hours of moderate physical work (based on heart rate). Heart rate and steps will be tracked whenever participants are wearing the watch, which is when they are awake. The watch is to be charged every night when they are sleeping. Participants will have to log down their physical activity by activating the physical activity tracker either on the watch or on the mobile application. If they did not hit the required level of physical activity, they will be sent a notification prompt through the mobile application with details of nearby workout locations as recommendation.
  Interventions: Device: Mobile phone application and smart watch
- Control Group (No Intervention): For the control group, they will wear the wearables as a tracking device for the period of the study (6 months). No prompts will be given and the mobile application will only be installed but not used for this group.

INTERVENTIONS:
Device: Mobile phone application and smart watch — Mobile phone application prompts
  Arms: Intervention Group

SUMMARY:
This study intends to determine if smart watches and mobile phone application prompts can complement physical activity as a preventive intervention by motivating participants to exercise, so as to improve their physical and cognitive outcomes.

The investigators hypothesize that technology will help increase engagement in physical activity for the intervention group relative to the control group and subsequently improve cognitive and physical outcomes.

DETAILED DESCRIPTION:
This study aims to explore the role of technology -- in the form of smart watches and mobile phone application -- in physical activity enhancement on cognitive frailty outcomes. Cognitive frailty is defined here as having both physical frailty and cognitive impairment but does not satisfy criteria for Major Neurocognitive Disorder. The investigators postulate that for older adults, such technology will help increase engagement in physical activity with subsequent improvement in cognitive and physical outcomes at follow up. This is with the aim of preventing this particular group from deteriorating to cognitive frailty because of the accompanying increased risk for adverse outcomes and morbidity.

This pilot study will be a randomized control trial with 2 treatment arms. Assessments will be done prior to and following the intervention period. During the period of intervention, the wearable will act as a tracking device and will be paired with a mobile application to issue prompts to the participant when necessary. The independent variable explored in the study is the use of the wearable while the levels of physical and cognitive improvements are the dependent measures. These will be tracked at baseline, 3 months and 6 months. Additionally, the mediating variable measured is the levels of physical activity to ensure that the proposed outcomes are affected through an increased level of physical activity encouraged by the use of the device.

If innovations like technology and the role of self-management proves efficacious, the future of healthcare in the context of a rapidly aging population will be more sustainable. Furthermore, this supporting role of technology in positive behavioral modification amongst older adults can have a multitude of applications in subsequent healthcare interventions.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 60 to 85 years

Exclusion Criteria:

* Engages in vigorous exercises as determined by having more than 0 minutes of vigorous exercise on the International Physical Activity Questionnaire (IPAQ).
* Has medical contraindications for exercising, including but not limited to: physical disabilities or heart conditions where the primary doctor disallows exercising at moderate intensity.
* Does not own an Android phone which can support at least a version 6.0 Operating System

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in frailty screening scores on the FRAIL questionnaire at 3 and 6 months | At 3 months and 6 months
  5 questions on fatigue, resistance, ambulation, illness and loss of weight. It is a simple screening test for frailty. Scores of 0 (non-frail), 1-2 (pre-frail) and 3-5 (frail).
Mean Change from Baseline in physical frailty as measured by physical performance tests at 3 months and 6 months | At 3 months and 6 months
  Hand grip strength in kilograms
Mean Change from Baseline in physical frailty as measured by physical performance tests at 3 months and 6 months | At 3 months and 6 months
  Gait speed, time taken to walk a specified distance as fast as possible, in seconds
Mean Change from Baseline in physical frailty as measured by physical performance tests at 3 months and 6 months | At 3 months and 6 months
  Timed Up and Go (TUG), time taken to stand up from a chair, walk 3 meters, turn around and sit back down, in seconds
Mean Change from Baseline in physical frailty as measured by physical performance tests at 3 months and 6 months | At 3 months and 6 months
  Chair Stand Test, time taken to stand up fully 5 times from a chair in seconds
Mean Change from Baseline in cognitive scores as measured on the Neurocognitive Assessment test battery at 3 and 6 months | At 3 months and 6 months
  Rey Auditory Verbal Learning Test (RAVLT) assesses verbal learning and memory
Mean Change from Baseline in cognitive scores as measured on the Neurocognitive Assessment test battery at 3 and 6 months | At 3 months and 6 months
  Digit Span Forward and Backward (DS) assesses working memory capacity
Mean Change from Baseline in cognitive scores as measured on the Neurocognitive Assessment test battery at 3 and 6 months | At 3 months and 6 months
  Colour Trails Test (CTT) assesses visual-spatial skills and attention
Mean Change from Baseline in cognitive scores as measured on the Neurocognitive Assessment test battery at 3 and 6 months | At 3 months and 6 months
  Wechsler's Block Design (WBS) assesses visuospatial ability
Mean Change from Baseline in cognitive scores as measured on the Neurocognitive Assessment test battery at 3 and 6 months | At 3 months and 6 months
  Semantic Fluency - animals (SFA) assesses semantic memory

SECONDARY OUTCOMES:
Mean Change from Baseline in Steps Taken measured by the smart watch at 3 months and 6 months | At 3 months and 6 months
  Number of steps taken daily
Mean Change from Baseline in moderate exercise measured by the smart watch at 3 months and 6 months | At 3 months and 6 months
  Minutes of moderate exercise in a week
Mean Change from Baseline in levels of physical activity measured by the "International Physical Activity Questionnaire" at 3 months and 6 months | At 3 months and 6 months
  Self-reported minutes and hours of vigorous or moderate exercise

OTHER OUTCOMES:
Control variable of sleep quality as measured on the Pittsburgh Sleep Quality Index (PSQI) at 3 and 6 months | At 3 months and 6 months
  Self-reported questionnaire on sleep quality in the last month. Global score ranges from 0-21 with a score of 5 and above indicating poor sleep quality. The higher the score, the poorer the sleep quality.
Control variable of levels of motivation as measured on the Barriers Self-efficacy Scale at 3 and 6 months | At 3 months and 6 months
  Self-reported questionnaire on levels of motivation specific to exercising. Scores ranges from 0-100. The higher the score, the higher the level of self-efficacy.
Control variable of depression as measured on the Geriatric Depression Scale at 3 and 6 months | At 3 months and 6 months
  Self-reported screening test for depression. Scores ranges from 0-15 and a higher score reflect more depressive symptoms.
Control variable of anxiety as measured on the Geriatric Anxiety Inventory at 3 and 6 months | At 3 months and 6 months
  Self-reported screening test for anxiety. Scores ranges from 0-20 and a higher score reflect more anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Rathi Mahendran, MMed (Psych), Principal Investigator — National University of Singapore
Locations (1):
- Hannah Senior Activity Center, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiah Hui Siew S, Yu J, Teo TL, Chua KC, Mahendran R, Rawtaer I. Technology and physical activity for preventing cognitive and physical decline in older adults: Protocol of a pilot RCT. PLoS One. 2024 Feb 23;19(2):e0293340. doi: 10.1371/journal.pone.0293340. eCollection 2024. PMID 38394113